CLINICAL TRIAL: NCT07169942
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Study Evaluating the Effects of Aleniglipron (GSBR-1290) on Body Composition in Participants Living With Obesity (Body Mass Index ≥ 30 kg/m2)
Brief Title: Aleniglipron Phase 2 Body Composition Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gasherbrum Bio, Inc., a wholly owned subsidiary of Structure Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GSBR-1290-16
Record Dates: First submitted 2025-08-20; First posted 2025-09-12 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Overweight, or Chronic Weight Management
Keywords: obesity, overweight, GSBR-1290, aleniglipron, chronic weight management, obese, small molecule, GLP-1 receptor agonist, body composition, Structure Therapeutics
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive aleniglipron or placebo administered orally.
  Interventions: Drug: aleniglipron or placebo
- Cohort 2 (Experimental): Participants will receive aleniglipron or placebo administered orally.
  Interventions: Drug: aleniglipron or placebo

INTERVENTIONS:
Drug: aleniglipron or placebo — Drug: aleniglipron administered orally Drug: placebo administered orally

SUMMARY:
This is a randomized, double-blind, placebo-controlled study evaluating the effects of aleniglipron on body composition in participants living with obesity. Participants will be randomized to aleniglipron or placebo in a ratio of 5:1. Participants will receive multiple ascending QD doses of aleniglipron or placebo in titration steps of 4 weeks duration for a total of 40 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Participants age ≥18 years and <80 years, with BMI ≥30 kg/m2
* Screening HbA1c <6.5 %

Exclusion Criteria:

* Previous documented diagnosis of diabetes mellitus
* Self-reported change in body weight >5% within 3 months before Screening
* Have a body weight, height, and/or width that prohibits the ability to obtain accurate measurements according to the DXA study specific manual that allows hemi-scan
* Have a prior or planned surgical treatment for obesity (excluding liposuction or abdominoplasty, if performed >1 year prior to screening)
* Have obesity induced by other endocrine disorders (such as Cushing's syndrome, Prader-Willi syndrome, or melanocortin 4 receptor deficiency)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 71 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percent change in total body fat mass by DXA | Baseline and week 40

SECONDARY OUTCOMES:
Percent change in visceral adipose tissue [VAT] by DXA | Baseline and week 40
Percent change in lean body mass by DXA | Baseline and week 40
Percent change in body weight by DXA | Baseline and week 40
Percent change in waist circumference | Baseline and week 40

OTHER OUTCOMES:
Change in patient-reported outcome SF-36 acute version | Baseline and week 40
Change in patient-reported outcome IWQOL-Lite CT | Baseline and week 40
Change in patient-reported outcome hunger/satiety evaluation checklist | Baseline and week 40
Change in high-density lipoprotein and low-density lipoprotein cholesterol | Baseline and week 40

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Research Site, Phoenix, Arizona
  - Research Site, Chicago, Illinois
  - Research Site, Richfield, Minnesota
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Rochester, New York
  - Research Site, Wilmington, North Carolina
  - Research Site, Norman, Oklahoma
  - Research Site, Moncks Corner, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Austin, Texas
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address a specific research question in an approved data sharing request
Supporting Information: Study Protocol
Time Frame: Data sharing requests will be considered beginning 36 months after the study publication (manuscript accepted for publication) and either 1) the product has been granted marketing authorization in at least two regulatory jurisdictions, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Researchers will submit a request containing the research objectives, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). Gasherbrum Bio, Inc. does not grant external requests for individual de-identified patient data for the following purposes:
  * Re-evaluating safety and efficacy end points already addressed in the product labelling,
  * Assessing safety or efficacy for an indication in current development Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a panel of external advisors. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement.